CLINICAL TRIAL: NCT03272256
Title: A Multi Center, Open-label, Phase 1 Clinical Trial to Evaluate the Safety, Tolerability, and Preliminary Efficacy of IM156 in Patients With Advanced Solid Tumors and Lymphoma
Brief Title: Phase 1 Study of IM156 in Patients With Advanced Solid Tumor and Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: ImmunoMet Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: IM_IM156-01
Record Dates: First submitted 2017-08-29; First posted 2017-09-05 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IM156, Dose escalation (Experimental)
  Interventions: Drug: IM156

INTERVENTIONS:
Drug: IM156 — Sequential 3+3 design.

SUMMARY:
The main purpose of first-in-human IM156 study is to evaluate the safety and tolerability, and to determine the maximum tolerated dose and recommended phase 2 dose of IM156.

ELIGIBILITY:
Inclusion Criteria:

1. Aged at least 19 years old.
2. Patients histologically or cytologically diagnosed with advanced solid tumor.
3. Patients for whom no standard therapies are available or who have failed in the existing conventional therapies.
4. Patients with a measurable or evaluable lesion by the RECIST v1.1 [for patients with recurrent glioblastoma, the RANO guideline is applied].
5. Patients with the Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2.
6. Patients with the adequate function of bone marrow, kidney and liver as follows.

   ① Absolute Neutrophil Count ≥ 1,500/mm³, Platelet ≥ 100,000/mm³, Hemoglobin ≥ 9.0 g/dL (In case of hemoglobin < 9.0 g/dL, the patient can be enrolled if the value is reversed to ≥ 9.0 g/dL. However, blood transfusion to meet this criterion within 1 week is not allowed.)

   ② Serum creatinine ≤ 1.5 X upper limit of normal (ULN)

   ③ Total bilirubin ≤ 1.5 X UNL, AST, ALT ≤ 3 ×ULN (for patients with liver disease ≤ 5 ×ULN)

   ④ Fasting serum glucose ≤ 160 mg/dL
7. Patients with the life expectancy ≥ 12 weeks.
8. Patients who have agreed to use acceptable methods for contraception during the study treatment period.

   (e.g.: sterilization of the patient and his/her partner, intrauterine device of the partner, barrier contraception, combination with diaphragm or condom)
9. Patients who have voluntarily signed an informed consent to participate in this clinical study.

Exclusion Criteria:

1. Patients with a history of hypersensitivity to the active ingredient or any component of the investigational product or biguanides.
2. Patients with a current evidence of diabetes mellitus who are currently being treated with another biguanide (e.g., metformin)
3. Patients with a history of serious gastrointestinal bleeding within 6 weeks prior to screening or patients with any disease possibly affecting the absorption of oral agents. (malabsorption syndrome, hemorrhagic gastric ulcer, etc.)
4. At the time of screening,

   * For patients who underwent major surgery, at least 4 weeks have not elapsed after surgery.
   * For patients who underwent radiotherapy, at least 3 weeks have not elapsed from the last treatment day.
   * For patients who underwent chemotherapy, at least 3 weeks have not elapsed from the last treatment day. (6 weeks for nitrosurea compounds).
   * For patients treated with biologic agents including hormone therapy, at least 5 half-lives or 3 weeks, whichever is shorter.
5. Patients who have not been recovered from the toxicities to grade 1 of the therapy received prior to screening.
6. Pregnant women or nursing mothers.
7. Patients who were administered another investigational product within 3 weeks prior to screening.
8. Patients with uncontrolled metastasis to the central nervous system. However, patients with treated and stable brain metastases (stable at least for 30 days on radiology imaging) are allowed to enroll.
9. Patients with suspected serious infectious diseases, intestinal paralysis, bowel obstruction, interstitial pneumonia, or pulmonary fibrosis.
10. Patients with a history of psychiatric disorders likely to threaten the compliance with this protocol.
11. Patients with a history of alcohol or drug abuse within 12 weeks prior to screening.
12. Human Immunodeficiency Virus (HIV) infection or active hepatitis B or C. Patients with no detectable viral load could be enrolled.
13. Patients with severe traumatism.
14. Patients with any clinically significant abnormal intestinal findings that may interfere with the administration, passage, or absorption of the investigational product, which makes the patients unable to orally take the tablet form of drugs.
15. Patients with severe cardiac disorders (e.g. myocardial infarction, congestive heart failure, arrhythmia showing dramatic change in electrocardiogram (ECG), severe or unstable angina, other serious cardiac disorders) or patients with comorbidities of other serious internal disorders (e.g. uncontrolled diabetes mellitus, chronic obstructive pulmonary disorder, renal failure, etc.) on investigator's judgment.
16. Patients who are otherwise considered to be ineligible for this study on investigator's judgment.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2019-12-02 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) | 4 weeks
  Evaluate the safety and tolerability to determine the maximum tolerated dose (MTD) and/or recommended phase 2 dose (RP2D)

SECONDARY OUTCOMES:
Maximum plasma concentration (Cmax) | 4 weeks
Time to Cmax (Tmax) | 4 weeks
Area under the curve (AUC) | 4 weeks
Plasma half life (T1/2) | 4 weeks
Volume of distribution (V/F) | 4 weeks
Plasma Clearance (CL/F) | 4 weeks
Exploratory Surrogate Biomarker | 2 weeks
  Explore potential surrogate biomarkers in peripheral blood mononuclear cells (PBMC).
Preliminary tumor response | Every 8 weeks up to end of treatment (EOT)
  Assess objective tumor response and progression based on the Response Evaluation Criteria for Solid Tumor (RECIST) v1.1 [for patients with recurrent glioblastoma, the Response Assessment in Neuro-Oncology (RANO) guideline is applied].

CONTACTS AND LOCATIONS:
Overall Officials: Sun Young Rha, MD, PhD, Principal Investigator — Department of oncology
Locations (3):
- South Korea (3):
  - CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do
  - Asan Medical Center, Seoul
  - Yonsei University Severance Hospital, Seoul